CLINICAL TRIAL: NCT07316569
Title: Healthy Eating and Active Living to Reverse Diabetes Pilot Study
Brief Title: The Healthy Eating and Active Living to Reverse Diabetes Pilot Study
Acronym: HEAL Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Principal Investigator, James E. Bailey, MD, MPH, Executive Director, Tennessee Population Health Consortium, University of Tennessee
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-09351-FB UM; A23-0844-001 (Other: UTHSC Office of Sponsored Programs)
Record Dates: First submitted 2025-12-02; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Diabete Type 2; Diabetes; Overweight , Obesity
Keywords: multicomponent; behavioral change; lifestyle; diet; weight loss; pragmatic; healthy eating; health coaching; community-based diabetes care
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Overweight; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Care (Active Comparator): Participants in this arm received enhanced usual care only. Enhanced usual care consisted of standard diabetes education, health coaching, and routine clinical management provided by their existing healthcare providers. No additional study-delivered classes, coaching, or materials were provided. Participants completed study assessments on the same schedule as the intervention group.
  Interventions: Behavioral: Enhanced Usual Diabetes Care
- Intensive Care (Multicomponent Intervention) (Experimental): Participants in this arm received a structured, multicomponent diabetes remission intervention promoting healthy eating and intensive weight loss in addition to usual care. The intervention included biweekly group sessions over the study period, covering nutrition and weight management; cooking classes; individual health coaching; 3-month diet replacement; and physician-supervised medication discontinuation. The program also included goal-setting, progress check-ins, and supportive accountability delivered by health coaches. Participants completed the same study assessments as the enhanced care arm.
  Interventions: Behavioral: Intensive Multicomponent Healthy Eating and Weight Loss Intervention

INTERVENTIONS:
Behavioral: Intensive Multicomponent Healthy Eating and Weight Loss Intervention — An intensive multicomponent diet and weight-loss intervention designed to support diabetes remission. The program included biweekly group sessions focused on low-carbohydrate, moderate-fat nutrition strategies; portion and calorie guidance; behavior-change skills; goal-setting; and weight-tracking. Participants also completed biweekly individual health-coaching sessions that provided personalized dietary guidance, problem-solving support, and adherence monitoring. The intervention incorporated 12 weeks of weekly total diet replacement provided through home delivery of lower-carbohydrate, lean-protein food items to facilitate adherence to dietary goals. During the total diet replacement phase participants also received physician-supervised medication discontinuation. Physical activity recommendations and strategies for managing blood glucose were also covered. The intervention was delivered by health coaches and provided in addition to participants' usual clinical care.
  Arms: Intensive Care (Multicomponent Intervention)
Behavioral: Enhanced Usual Diabetes Care — Participants received enhanced usual diabetes care. This included optional diabetes self-management education provided through routine clinic services, individualized health-coaching sessions provided at neighborhood health hub facilities focused on general diabetes management support. In addition, participants received four produce vouchers valued at $50 each to promote access to fresh fruits and vegetables. No additional study-delivered classes, dietary programming, or supplemental food items were provided.
  Arms: Enhanced Care

SUMMARY:
The HEAL Diabetes Program is a multicomponent intensive plant-forward healthy eating program designed to reverse diabetes. Several recent studies, most notably the Diabetes UK-funded Diabetes Remission Clinical Trial (DiRECT) in England and Scotland, have demonstrated that intensive programs for weight loss and weight loss maintenance can lead to long-term remission of diabetes for as many as half of patients with early Type 2 (adult-onset) diabetes. Furthermore, the U.S. Preventive Services Task Force has recommended that all patients with obesity and at highest risk for diabetes be referred to such intensive multicomponent behavioral weight loss interventions, but no such programs are available for people living in the low-income and underserved areas of Memphis. This effort will pilot an innovative, culturally tailored, and intensive healthy eating program designed to reverse diabetes based in the UTHSC Neighborhood Health Hub located in low-income neighborhoods to demonstrate that this approach will work in Memphis to improve and extend people's lives. The HEAL Diabetes Pilot Program will: a) engage and retain a minimum of 30 patients with Type 2 diabetes and obesity to participate in the program as well as 30 additional "control" patients who will receive routine care, and b) assess patient outcomes including weight loss and rates of diabetes remission using average blood sugar (hemoglobin A1c) over a six-month period. The healthy eating and active living to reverse diabetes (HEAL Diabetes) is a pilot study that aims to evaluate the feasibility, effectiveness, and operational and financial sustainability of a multicomponent health coach-supported nutrition intervention in a predominately African American population in Memphis, Tennessee. The investigators aim to assess study feasibility by evaluating recruitment, sample characteristics, intervention acceptability and procedural suitability. The investigators also aim to quantify and compare the treatment and control groups on primary outcomes including changes in body weight, hemoglobin A1c (HbA1c), and proportion of patients who achieved diabetes remission (HbA1c25 < 6.5%) from baseline to 12-months. Additionally, the investigators aim to assess changes in diabetes self-efficacy and self-care activities and examine cost effectiveness of the multicomponent intervention. Drawing on evidence from DiRECT, MODEL, and related studies, the investigators hypothesize that the intervention arm will achieve greater weight loss and higher diabetes remission than the control. Additionally, the investigators hypothesize that the program will be operationally and financially sustainable.

ELIGIBILITY:
Inclusion Criteria: Patients must meet the following criteria to be eligible:

* adults 18 years or older
* a type 2 diabetes (T2D) duration of 0-6 years (diagnosis based on one recorded HbA1c test)
* HbA1c value ≥ 6.5 percent at the screening visit
* BMI ≥ 25 kg/m2
* access to a cell phone or smartphone with texting and voicemail capabilities

Exclusion Criteria:

* current use of insulin or more than two hypoglycemic medications (either oral or injectable)
* a recent routine HbA1c greater than or equal to 12%
* weight loss of >5 kg within the last six months
* inability to understand consent procedures, understand and speak English
* pregnancy or considering pregnancy
* diagnosis or exhibited unstable psychiatric condition, dementia, neurological disorder, or history of severe head trauma or brain tumor, and cognitive impairment
* perceived unwillingness or inability to participate
* planned move from the region during the study
* participation in another clinical research trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-10-11 (Actual); Primary Completion 2025-08-02 (Actual); Study Completion 2025-08-02 (Actual)

PRIMARY OUTCOMES:
Change in Body Weight | From enrollment to the end of 6 months.
  Change in body weight in pounds from baseline to 6 months
Change in Hemoglobin A1c (HbA1c) | Baseline to 6 months
  Change in HbA1c (%) from baseline to 6 months
Proportion of Participants Achieving Diabetes Remission | 6 months
  Proportion of participants achieving diabetes remission at 6 months, defined as HbA1c < 6.5% without use of glucose-lowering medications for at least 2 months

SECONDARY OUTCOMES:
Change in Random Blood Glucose | Baseline to 6 months
  Change in random (non-fasting) blood glucose concentration from baseline to 6 months, measured using standard capillary or venous blood glucose testing in Milligrams per deciliter (mg/dL).
Change in Diabetes Self-Efficacy Score | Baseline to 6 months
  Change in diabetes self-efficacy from baseline to 6 months, assessed using the Stanford Diabetes Self-Efficacy Scale (DSES).
Change in Diabetes Self-Care Activities Score | Baseline to 6 months
  Change in diabetes self-care behaviors from baseline to 6 months, assessed using the Summary of Diabetes Self-Care Activities (SDSCA).
Cost of Intervention Delivery | 6 months
  Total cost of delivering the intervention over 6 months, including personnel, materials, and program implementation expenses, estimated to inform potential scalability of the intervention.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UTHSC Health Hub-Uptown, Memphis, Tennessee
  - UTHSC Health Hub-ShelbyCares, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset contains sensitive, identifiable health information, and sharing could compromise participant privacy. Data are intended for use only by the study team for the purposes outlined in the study protocol.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT07316569/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT07316569/ICF_001.pdf